CLINICAL TRIAL: NCT02540382
Title: Comparison of Covered and Bare Stent in TIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Liu Fuquan, Department of Interventional Therapy, Beijing Shijitan Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: liufq_sjt
Record Dates: First submitted 2015-08-27; First posted 2015-09-03 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Cirrhosis
Keywords: TIPS; Hepatocellular Carcinoma; Portasystemic Shunt
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- covered stent (Experimental): Procedure/Surgery: Jugular vein puncture and catheterization. Device: RUPS-100 (COOK Company) sheath, 8 mm balloon, Pigtail catheter, 8 mm covered stents (Bard, Fluency).
  Drug (including placebo): No Biological/Vaccine: No Radiation: No Behavioral (e.g., Psychotherapy, Lifestyle Counseling): No Genetic (including gene transfer, stem cell and recombinant DNA): No Dietary Supplement (e.g., vitamins, minerals): No.
  Interventions: Device: covered stent
- bare stent (Other): Surgery: Jugular vein puncture and catheterization. Device: RUPS-100 (COOK Company) sheath, 8 mm balloon, Pigtail catheter, 8 mm bare stents (EV3, protégé; Cordis, Smart).
  Drug (including placebo): No Biological/Vaccine: No Radiation: No Behavioral (e.g., Psychotherapy, Lifestyle Counseling): No Genetic (including gene transfer, stem cell and recombinant DNA): No Dietary Supplement (e.g., vitamins, minerals): No.
  Interventions: Device: bare stent

INTERVENTIONS:
Device: covered stent — A broad range of implant diameters and lengths for the treatment of in-stent restenotic peripheral and central lesions* in patients with AV grafts and AV fistulae Small incremental stent graft lengths to help maintain venous real estate and cannulation area Minimal shortening and radiopaque markers aid in excellent placement accuracy
  Arms: covered stent
Device: bare stent — A one piece laser cut, self-expanding nitinol stent combining a micromesh design with a multi segmental construction.
  The 36 strut, 6 bridge construction of the Stent provides an unmatched balance of radial force, scaffolding, and longitudinal stability.
  The design offers crush recoverable flexibility in the most challenging vasculature, with optimal wall apposition, conformability and minimal foreshortening.
  It offers a broad portfolio of sizes for the treatment of routine and challenging Iliofemoral lesions.
  Arms: bare stent

SUMMARY:
Investigators aim to compare the efficacy of 8 mm Fluency covered stent and bare stent in transjugular intrahepatic portosystemic shunt (TIPS) for the treatment of cirrhotic portal hypertension.

DETAILED DESCRIPTION:
From January 2006 to December 2010, the covered (experimental group) or bare stent (control group) was used in 131 and 127 patients, respectively. The recurrence rates of gastrointestinal bleeding and refractory hydrothorax/ascites, the cumulative restenosis rates in 1, 2, 3, 4, and 5-years, the incidence rate of hepatic encephalopathy, the rate of secondary interventional therapy, the 1, 2, 3, 4 and 5-year survival rates were compared between the experimental group and the control group.

ELIGIBILITY:
Inclusion Criteria:

1. portal hypertension patients with defined indications for TIPS treatment;
2. scheduled for elective TIPS; and
3. aged between 18-70 years.

Exclusion Criteria:

1. combined with hepatic encephalopathy before the treatment;
2. combined with portal vein thrombosis;
3. combined with malignant liver tumor or malignancies at the other sites; or
4. combined with hemorrhage of gastrointestinal ulcer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2006-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
restenosis/occlusion rate | up to 5 years
  The cumulative restenosis rate in 1, 2, 3, 4, or 5-year

SECONDARY OUTCOMES:
recurrence rate of gastrointestinal bleeding | up to 5 years
recurrence rate of refractory hydrothorax/ascites | up to 5 years
  the recurrence rate of refractory hydrothorax/ascites (including non-responders, recurrent, and newly developed cases) during the follow up
survival rate | up to 5 years
  The 1, 2, 3, 4 and 5-year survival rate
rate of secondary interventional therapy | up to 5 years
  rate of secondary interventional therapy
incidence rate of hepatic encephalopathy | up to 5 years
  The incidence rate of hepatic encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Jianli Xu, MD, PhD, Study Chair — Beijing Shijitan Hospital, Capital Medical University
Locations (1):
- Beijing Shijitan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li HB, Yue ZD, Zhao HW, Wang L, Fan ZH, He FL, Dong XQ, Liu FQ. Pathological Features of Mitochondrial Ultrastructure Predict Susceptibility to Post-TIPS Hepatic Encephalopathy. Can J Gastroenterol Hepatol. 2018 Jul 16;2018:4671590. doi: 10.1155/2018/4671590. eCollection 2018. PMID 30079331